CLINICAL TRIAL: NCT04181255
Title: The Cold Heart Study: A Randomized Pilot Trial of Surfactant Therapy Following Deep Hypothermic Circulatory Arrest During Cardiac Surgery
Brief Title: Cold Heart Study: A Randomized Pilot Trial of Surfactant Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator Retirement
Sponsor: University of Michigan (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Steven Donn, M.D., Professor Emeritus of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00160492
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Congenital Heart Disease; Hypoplastic Left Heart Syndrome
Keywords: Norwood procedure
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome | interventions — poractant alfa; Surface-Active Agents; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curosurf (Experimental)
  Interventions: Drug: Curosurf
- Sham (air) (Placebo Comparator)
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Curosurf — This arm will consist of a single dose of Curosurf (200 mg/kg) that will be given in the Pediatric Cardiothoracic Unit (PCTU) after surgery once the subject has reached a normalized body temperature.
  Other Names: poractant alfa; surfactant
  Arms: Curosurf
Drug: Sham — This arm will consist of a single dose of sham (air) that will be given through the endotracheal tube in the Pediatric Cardiothoracic Intensive Care Unit after surgery once the subject has reached a normalized body temperature.
  Arms: Sham (air)

SUMMARY:
This clinical trial is being done to see if giving surfactant (Curosurf®) will decrease the number of days that infants will need a breathing tube, decrease the days in the critical care unit and decrease the number of days needed in the hospital. The primary hypothesis for this study is that there will be fewer days needed on mechanical ventilation and improved lung compliance and pulmonary gas exchange.

DETAILED DESCRIPTION:
This study will enroll infants undergoing cardiothoracic surgery requiring deep hypothermic circulatory arrest (DHCA) at the University of Michigan's C.S. Mott Children's Hospital. Patients that are eligible will be randomized to receive either one dose surfactant or the sham (air) arm after the surgical procedure. Patients will be monitored for an additional 30 days after the breathing tube is removed. It is possible that subjects may be discharged prior to the last assessment, therefore for subjects who have been discharged a member of the study team will contact the parent (s) or legal authorized representative by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than or equal to 12 weeks of age with hypoplastic left heart syndrome (HLHS) undergoing cardiothoracic surgical correction (Norwood) requiring DHCA.
* Infants weighing 2500 grams or greater at the time of surgery.
* Written informed consent from parent(s) or legally appointed representative (LAR).

Exclusion Criteria:

* Patients who are less than 36 weeks Post Menstrual Age (PMA) at the time of surgical correction.
* Underlying craniofacial, airway or lung anomalies which could compromise administration of surfactant.
* Infants weighing less than 2500 grams at the time of the surgical correction.
* Mechanical ventilation for> 7 days prior to surgical correction.

Ages: 1 Day to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Number of days of mechanical ventilation | Throughout hospitalization (approximate average 5 days)
  This will be the number of days from intubation to the extubation date.
Number of days in the Pediatric Cardiothoracic Unit | Approximately 11 days
  From time of admission until transfer out of the unit.
Number of post-operative hospital days | Up to 1 year

SECONDARY OUTCOMES:
Total number of patients requiring thoracostomy tube placement for air leak not associated with standard post-operative management prior to extubation | Approximately 1 week
  Post-surgery prior to extubation.
Total number of patients requiring high frequency ventilation (HFV) (High frequency oscillator ventilation or High frequency jet ventilation) | Up to 1 year
  Post-surgery throughout hospitalization.
Total number of patients requiring extracorporeal membrane oxygenation (ECMO) for pulmonary failure | Up to 1 year
  Post-surgery throughout hospitalization.
Changes in positive end-expiratory pressures post intervention | Baseline to approximately 1 week
  After therapy until extubation.
Changes in peak inspiratory pressures post intervention | Baseline to approximately 1 week
  After therapy until extubation.
Changes in dynamic lung compliance post intervention | Baseline to approximately 1 week
  After therapy until extubation.
Changes in oxygen requirements post intervention | Baseline to approximately 1 week
  After therapy until extubation.
Changes in oxygenation index (OI) post intervention | Baseline to approximately 1 week
  OI is the product of mean airway pressure and fraction of inspired oxygen divided by the partial pressure of oxygen. After therapy until extubation.
Time to successful extubation readiness trials (ERT) post intervention | Approximately 1 week
  Measured in hours until successful ERT, and then successful extubation. Not everyone who passes an ERT is immediately extubated (typically done once per day), so the plan is daily.
  Successful extubation is defined as remaining extubated for 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Donn, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No